CLINICAL TRIAL: NCT07343271
Title: Dual-energy CT vs. MRI in the Evaluation of Squamous Cell Carcinomas of the Oral Cavity and Oropharynx
Acronym: DECT-CEco
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9773
Record Dates: First submitted 2026-01-06; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Oral Squamous Cell Carcinoma; Oropharyngeal Squamous Cell Carcinoma
Keywords: Oral Squamous Cell Carcinoma; Oropharyngeal Squamous Cell Carcinoma; TNM stage of the tumor
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The diagnostic and pre-therapeutic assessment of squamous cell carcinomas requires a neck and chest CT scan and a neck and facial MRI, which is the most effective examination, to establish the TNM stage of the tumor. However, obtaining this complete assessment can delay treatment. Confirmation of the non-inferiority of 40keV dual-energy CT in BOLT compared to MRI would spare the patient an additional MRI examination, speed up the pre-treatment assessment, reduce the loss of opportunity due to delayed treatment, and free up MRI imaging slots, which are still insufficient in the region.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (≥18 years)
* presenting with oral or oropharyngeal squamous cell carcinoma proven by histopathological analysis of a biopsy
* having undergone a clinical examination with nasofibroscopy by an ENT surgeon specializing in cancer surgery
* a contrast-enhanced cervicofacial MRI
* and a contrast-enhanced cervicofacial DECT with BOLT maneuver.

Exclusion Criteria:

* A lesion other than oral or oropharyngeal squamous cell carcinoma
* A labial location
* A contraindication to performing one or both of the imaging examinations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patient presenting with oral or oropharyngeal squamous cell carcinoma proven by histopathological analysis of a biopsy
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-07-11 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07-11 (Estimated)

PRIMARY OUTCOMES:
Overall agreement established by interclass correlation on the T stage of TNM | Up to 12 months
  Overall agreement established by interclass correlation on the T stage of TNM between the radiological analysis of the DECT 40 kev BOLT, and of the MRI, compared to the reference T stage of TNM from the RCP:
  Overall agreement:
  This means: do the methods give the same results? We want to know if DECT and MRI reach the same T stage for the same patient.
  Example:
  DECT: T3 MRI: T3 Result: Good agreement
  DECT: T2 MRI: T3 Result: Disagreement

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'ORL et de Chirurgie Cervico-faciale - CHU de Strasbourg - France, Strasbourg, France